CLINICAL TRIAL: NCT02502461
Title: Tracheal Palpation of Sliding Cuff to Assess Endotracheal Tube Location in Trachea - A Randomized Controlled Trial
Brief Title: Tracheal Palpation of Sliding Cuff to Assess Endotracheal Tube Location
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, William McKay, Professor of Anesthesia, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Bio#15-63
Record Dates: First submitted 2015-07-13; First posted 2015-07-20 (Estimated); Results first posted 2019-03-06 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2018-11

CONDITIONS: Anesthesia Intubation Complication

STUDY DESIGN:
Intervention Model Description: Double-blind RCT
Who Masked: Participant, Outcomes Assessor
Masking Description: Participant is fully anesthetized. 1)Depth of ETT not known or knowable until after objective measurement. 2) Pain assessor unaware of participant group.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- standard care (Sham Comparator): Intervention: Subject intubated in routine fashion by the attending anesthesiologist with cuffed endotracheal tube; endotracheal tube cuff inflated; tube taped in place; depth measured bronchoscopically; patient asked to rate soreness of throat on verbal response scale when awake postoperatively.
  Interventions: Procedure: cuff palpation
- cuff palpation (Active Comparator): Intervention: Subject intubated in routine fashion by the attending anesthesiologist with cuffed endotracheal tube; endotracheal tube cuff inflated; inflated cuff palpated and depth adjusted accordingly; tube taped in place; depth measured bronchoscopically; patient asked to rate soreness of throat on verbal response scale when awake postoperatively.
  Interventions: Procedure: cuff palpation

INTERVENTIONS:
Procedure: cuff palpation — Inflated endotracheal tube cuff palpated through anterior extra-thoracic trachea while tube is gently moved to place the cuff midway between cricoid and sternal notch.

SUMMARY:
Correct endotracheal tube (ETT) placement is important. Proper ETT position is achieved when the distal tip is in mid-trachea with the head in neutral alignment. Unrecognized tube misplacement is an uncommon but significant cause of hypoxemia and death during general anesthesia as well as in the care of critically ill patients.

Hypotheses: A specific manoeuvre to palpate the inflated ETT cuff, with fingers anterior to the trachea, moving the ETT caudally then rostrally following intubation, will enable correct depth placement of the tip of the ETT within the trachea (more than 2.5cm above the carina with cuff below the vocal cords) more frequently than routine care. This will not cause tissue damage as measured by sore throat.

DETAILED DESCRIPTION:
Introduction:

Correct endotracheal tube (ETT) placement is important. Proper ETT position is achieved when the distal tip is in mid-trachea with the head in neutral alignment. Unrecognized tube misplacement is an uncommon but significant cause of hypoxemia and death during general anesthesia as well as in the care of critically ill patients.

Three types of malpositioning can occur: one outside the trachea (esophageal), and two within the trachea: too shallow, or too deep (endobronchial). Esophageal intubation results in hypoxemia and inflation of the stomach. Too-shallow placement of the ETT can result in inadvertent extubation, especially with manipulation of head and neck. Endobronchial intubation occurs when the ETT is advanced into a mainstem bronchus, which results in hypoxia and the potential for barotrauma in the hyperventilated lung.

Confirmation of correct ETT placement is currently performed by several methods. In the operating room, simple measurement of the length of the tube at the corner of the mouth using marks on the ETT is the usual method (Measurement Method: MM; 21cm at the teeth for women; 23cm for men). It is simple and rapid, but not reliable. One study attempted to improve on this by using anatomical landmarks to determine ETT tube length as measured at the mouth. It enabled a reduction in the incidence of too-deep placement of the ETT from 58.8% to 24%. Measurement of these landmarks is sufficiently inconvenient that it is not widely practised.

Cuff ballottement at the level of the suprasternal notch is a technique that has been studied with cuffed tubes in adults. Ballottement involves moving the fingers in a radial axis of the ETT in order to compress and release the cuff, while feeling and watching the corresponding movement of the pilot balloon. Studies to date of ballottement do not comment on its ability to prevent esophageal intubation.

The investigators propose to refine methods of palpating the trachea which the investigators studied in a previous experiment. The investigators found that palpation of the anterior trachea with the fingertips enabled us to feel the tip of the endotracheal tube sliding into the trachea. That study showed that palpation of the trachea could enable correct position of the endotracheal tube with respect to depth.

The investigators have refined the manoeuvre and found a technique that deserves further study to assess whether it can determine tracheal depth. The investigators completed a small (N =30) pilot study of intubation of the trachea (manuscript in preparation), in which investigators palpate over the trachea in the anterior neck to feel the inflated cuff movement while the ETT is moved caudally, then rostrally (described in detail in "Procedures"). The investigator attempted to determine the depth of the endotracheal tube by feeling the cuff move under his fingers in the trachea. The endotracheal tube was then immobilized at that depth, and fibre-optic bronchoscopy used to determine depth of the tip in the trachea. That study showed that the technique was safe and resulted in only one ETT tip of 31 (3.2%) lying too close to the carina (<2.5cm) compared to 4 of 30 (15.4%) in the initial placement (difference not significant). It enabled some refinement with practice. Because the technique involves moving the ETT up and down in the trachea, it may cause irritation of the mucosa and pain. The investigators had no complaints from patients or reports of sore throat from PACU nurses in the pilot study, but did not specifically study that outcome. The present study is a Randomized Controlled Trial (RCT) with ETT correct depth as principal and sore throats as secondary endpoint.

Objectives

1. Primary outcome. To tabulate the incidence and severity of sore throat.
2. Secondary outcome.To tabulate the incidence and severity of sore throat.To assess the reliability of palpation of the sliding cuff as a method to determine depth of ETT in the trachea.

Hypotheses A specific manoeuvre to palpate the inflated ETT cuff, with fingers anterior to the trachea, moving the ETT caudally then rostrally following intubation, will enable correct depth placement of the tip of the ETT within the trachea (more than 2.5cm above the carina with cuff below the vocal cords) more frequently than routine care and will not cause tracheal damage as assessed by throat pain.

Patient safety Risk from moving the ETT with the cuff inflated is not precisely known. However, one of the investigators (WPM) has employed the technique routinely for 20 years in several thousand intubations with no apparent harmful effects.

Risk from gentle palpation of an anesthetized patient's neck with clean physician's fingers is negligible, as reported in the ballottement literature cited above.

Risks of fibre-optic bronchoscopy are, in general, very small. This is borne out by the limited literature; a review in English from 1988, and a recent review in Italian. Both describe rare complications from fibre-optic bronchoscopy only when biopsies are taken. There are no reported complications for fibre-optic bronchoscopy down an in situ endotracheal tube only to the depth of the carina in adults.

Clinical Utility If this technique proves safe and reliable, it can decrease the risk of ETT misplacement. Further, if it is reliable, it is clinically very useful because it takes no special equipment, it can be performed in less than 5 seconds in any intubating situation (from operating room to battlefield), and it may make x-ray confirmation unnecessary, avoiding radiation and expense.

Methods Subjects: Following University of Saskatchewan Research Ethics Board and Saskatoon Health Region approval, informed consent will be obtained from 90 subjects. The collection, use and disclosure of patients' private information will conform to the Health Information Protection Act (HIPA).

Randomization: Subjects will be randomized, only after intubation to ensure concealment, to a Cuff Palpation (CP) group or a No Palpation (NP) group. A numbered opaque envelope containing the assigned allocation will be opened. Blinding is not possible during intubation in this experiment, but the bronchoscopic measurement technique is not subjective. Assessment of throat pain in the post anesthetic care unit (PACU) will be by a blinded observer.

Measurements: Data will be recorded on paper data sheets for later transcription to a computer spread sheet for analysis. Usual demographics (age, gender, height, weight, type of surgery) will be recorded. The certainty of palpating the ETT cuff movement will be recorded (can/can't feel the cuff move), as will ETT depth at the teeth and bronchoscopically measured ETT depth in the trachea.

Experimental Intervention: Intubation will be by the attending anesthesiologist, who will choose the anesthetic, equipment, and intubating technique on clinical grounds. The anesthesiologists will be instructed to advance the tube to the depth of their choice. The cuff will be inflated to a measured pressure of 30cm water pressure, using a commercially available factory-calibrated device. After intubation, the patient's head will be placed resting on a small pillow in neutral position, and the patient will be randomized to CP or NP.

If CP, after the cuff is inflated, an investigator will palpate the trachea while advancing the ETT another 2 cm. If the cuff movement is not felt, the investigator will slowly withdraw the ETT until the cuff is palpated midway between the cricothyroid membrane and the sternal notch, where it will be fixed in place and its depth measured bronchoscopically. If NP, the cuff will be inflated, the ETT fixed in place, and the depth measured.

Once in place in the trachea, in both groups, the ETT will be moved carefully to the midline of the mouth without changing its tracheal depth, and the ETT depth marking at the upper incisors or gums noted. The ETT will be taped in place, and held by hand in place at that exact depth during bronchoscopy. Bronchoscopy will be carried out through the ETT via a bronchoscopic elbow connector, thus requiring no break in ventilation.

Depth of the ETT in the trachea will be determined by advancing the bronchoscope to just touch the carina, and the depth at the elbow connector marked with a spring clip applied to the bronchoscope. It will then be withdrawn to the ETT tip, and a second clip placed. The bronchoscope will be withdrawn further until the light glowing transmitted from the bronchoscope tip shines through the cricothyroid membrane, and a third clip placed on the bronchoscope. The bronchoscope will be removed and surgery will proceed. Measurements will be made of the distance between the clips.

Patients will be followed in PACU and asked to rate their throat pain using a validated 11 point numerical rating scale (NRS) for pain, where 0 is no pain, and 10 is the worst possible pain.

Statistical Analysis: Sample size for the primary outcome was calculated from the pilot study cited above that specified N = 88. The investigators will recruit 90 subjects to account for protocol violations. Sample size calculation for the pain of intubation assuming a difference of 2 with SD = 2 on a validated 11-point Verbal Response Scale (0 to 10) specifies 17 per group, or N = 34.

Demographics and frequency of cuff movement being palpable (P) or not palpable (N) will be reported. Actual depth of placement of ETT as confirmed by bronchoscopy will be reported by categories: "ETT too shallow" (part of cuff in vocal cords); "ETT too deep" (tip <2.5cm above carina); and "ETT placement satisfactory" (between those extremes), as described previously.18 Incidence of correct and incorrect placement will be compared between groups using Fisher's Exact test or Chi-squared. Intent-to-treat analysis will be used. Pain scores will be compared by independent-sample T-test.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) Class I and II patients
* ≥18 years of age
* undergoing elective surgical procedures in the Saskatoon acute care hospitals of the Saskatoon Health Region
* requiring endotracheal intubation as a component of the anesthetic plan.

Exclusion Criteria:

* those who are physiologically unstable
* when there is urgency to proceed with surgery
* patients requiring rapid sequence induction
* those with respiratory distress
* those for whom the attending anaesthesiologist feels it would compromise safety for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-07; Primary Completion 2016-07 (Actual); Study Completion 2016-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William P McKay, MD, Principal Investigator — University of Saskatchewan
Locations (1):
- Saskatoon Health Region, 410 22nd Street East, Saskatoon, Saskatchewan, Canada

REFERENCES:
- [Background] Owen RL, Cheney FW. Endobronchial intubation: a preventable complication. Anesthesiology. 1987 Aug;67(2):255-7. doi: 10.1097/00000542-198708000-00019. No abstract available. PMID 3605754
- [Background] Pollard RJ, Lobato EB. Endotracheal tube location verified reliably by cuff palpation. Anesth Analg. 1995 Jul;81(1):135-8. doi: 10.1097/00000539-199507000-00027. PMID 7598242
- [Result] McKay WP, Klonarakis J, Pelivanov V, O'Brien JM, Plewes C. Tracheal palpation to assess endotracheal tube depth: an exploratory study. Can J Anaesth. 2014 Mar;61(3):229-34. doi: 10.1007/s12630-013-0079-4. Epub 2013 Nov 21. PMID 24259250

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Care | Cuff Palpation
Started | 46 | 44
Completed | 46 | 44
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Care | Cuff Palpation | Total
Number analyzed (Participants) | 46 | 44 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (16) | 56 (16) | 56 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 28 | 51
  Male | 23 | 16 | 39

OUTCOME MEASURES:

1. Primary Outcome: Sore Throat
Description: Surrogate measure of tissue damage from moving the tube with cuff inflated = soreness of throat on an 11-point verbal pain scale, with 0 = no pain, and 10 the worst pain imaginable.
Time Frame: when patient awake (within 24 hours of intubation)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Care | Cuff Palpation
Number analyzed (Participants) | 46 | 44
units on a scale | 1.5 (2.1) | 0.6 (1.6)
Statistical Analysis 1: Comparison: Standard Care vs Cuff Palpation; Test type: Superiority; p = 0.04, t-test, 2 sided — Bonferroni correction; Mean Difference (Final Values) = 0.9, 95% CI 2-sided [0.1 to 1.7]

2. Secondary Outcome: Number of Participants With Correct Depth of Endotracheal Tube in Trachea,
Description: Endotracheal tube tip >2.5cm from carina and >5.5cm from vocal cords for women and >6cm from vocal cords for men
Time Frame: immediate (within 5minutes of intubation).
Population: Participants removed from analysis were all removed because of unavailable clean bronchoscope.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care | Cuff Palpation
Number analyzed (Participants) | 46 | 44
Participants | 19 | 29

ADVERSE EVENTS:
Arm/Group | Standard Care | Cuff Palpation
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/44
Other Adverse Events (participants affected / at risk) | 0/46 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes